CLINICAL TRIAL: NCT05094089
Title: Assessment of GORE® SYNECOR Biomaterial in Focused Patient Populations and Long-Term Application
Acronym: SYN 20-01
Status: Active, not recruiting | Type: Observational
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Other Study IDs: SYN 20-01
Record Dates: First submitted 2021-10-05; First posted 2021-10-26 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Hernia, Ventral; Hernia Incisional; Hernia Incisional Ventral
Keywords: Hernia Repair; Hernia Mesh Treatment; Ventral Hernia; Incisional Hernia; Intraperitoneal; Preperitoneal
MeSH Terms: conditions — Hernia, Ventral; Incisional Hernia | interventions — Herniorrhaphy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- SYNECOR IP Device: Hernia mesh repair with GORE® SYNECOR Intraperitoneal Biomaterial
  Interventions: Device: Hernia repair with mesh
- SYNECOR PRE Device: Hernia mesh repair with GORE® SYNECOR Preperitoneal Biomaterial
  Interventions: Device: Hernia repair with mesh

INTERVENTIONS:
Device: Hernia repair with mesh — Hernia repair with GORE® SYNECOR Biomaterial; technical approach laparoscopic, robotic or open surgical / minimally invasive surgery

SUMMARY:
The SYN 20-01 Study is a non-interventional, prospective, multicenter, multicohort, international, post-market clinical investigation looking into the assessment of GORE® SYNECOR Biomaterial in focused patient populations and in long-term application.

Patients with ventral / incisional hernia amenable to hernia mesh repair will be enrolled into two cohorts (US and EU cohort) and followed-up over the period of 60 months.

ELIGIBILITY:
Key Inclusion Criteria - IP Cohort:

* De-Novo ventral/incisional hernia amenable to repair with GORE® SYNECOR IP Biomaterial
* Clean wound (CDC Wound Class I)
* mVHWG Grade 1 or 2 (modified Ventral Hernia Working Group)

Key Exclusion Criteria - IP Cohort:

- Wound is either clean-contaminated, contaminated or dirty-infected

Key Inclusion Criteria - PRE Cohort:

* De-novo ventral/incisional hernia, with subject anatomy and surgical plan amenable to open surgical repair or minimally invasive surgery with the GORE® SYNECOR PRE Biomaterial placed in a sublay fashion within the preperitoneal space
* Clean wound (CDC Wound Class I)
* mVHWG Grade 1 or 2 (modified Ventral Hernia Working Group)

Key Exclusion Criteria - PRE Cohort:

- Wound is either clean-contaminated, contaminated or dirty-infected

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The SYN 20-01 study population will consist of patients who present with ventral/incisional hernia disease requiring treatment per the evaluating physician. Eligible study subjects need to be amenable to treatment with a permanent synthetic mesh as suggested by the inclusion and exclusion criteria for each study cohort.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2023-02-24 (Actual); Primary Completion 2030-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Hernia Recurrence | 24 Months
  Hernia Recurrence Treated Location
Hernia Recurrence | 60 Months
  Hernia Recurrence Treated Location

SECONDARY OUTCOMES:
Hospital Re-Admission | 60 Months
  Device or procedural-related
Thirty-Day Mortality | 30 Day
  Mortality of all causes
SSO within 24 months post-procedure | 24 Months
  Surgical Site Occurrence (SSO)
SSI (Surgical Site Infection) | 60 Months
  Surgical Site Infection (SSI)
Freedom from mesh-involved events | 60 Months
  Freedom from mesh-involved events
Major Seroma (clinically confirmed) | 60 Months
  Major Seroma as clinically assessed (physiological parameters) and defined as seroma requiring treatment in the presence of infection, recurrence, mesh rejection or the need to be punctured/aspirated will be described without specific hypothesis or formal goal. Number of subjects with reported major seroma will be described as clinically confirmed by the investigator.
Change in Quality of Life (QoL) - SF 36 Questionnaire | 60 Months
  SF 36 Questionnaire (36-Item Short Form Survey Instrument; possible score ranges from 0 to 100 points. 0 points represent the greatest possible limitation of health, while 100 points represent the absence of health restrictions)
Change in Quality of Life (QoL) - Carolinas Comfort Scale (CCS) | 60 Months
  Carolinas Comfort Scale (CCS); CCS was designed that a lower score indicates a favorable health status; the total score is based on a scale of 0 - 115)
Ventral Hernia Recurrence Inventory sensitivity / specificity within 60 Month Follow-Up | 60 Months
  VHRI Survey (Ventral Hernia Recurrence Inventory)
Adverse Events by Clavien Dindo Classification | 60 Months
  Adverse Events by Clavien Dindo Classification
Surgical Site Occurrences (SSOPI) requiring Procedural Intervention | 24 Months
  Surgical Site Occurrences (SSOPI) requiring Procedural Intervention
Surgical Site Occurrences (SSOPI) requiring Procedural Intervention | 60 Months
  Surgical Site Occurrences (SSOPI) requiring Procedural Intervention

CONTACTS AND LOCATIONS:
Locations (15):
- United States (8):
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Tufts Medical Center, Boston, Massachusetts
  - Corewell Health, Grand Rapids, Michigan
  - Lovelace Women's Hospital, Albuquerque, New Mexico
  - Stony Brook University Hospital, Stony Brook, New York
  - Novant Health New Hanover Regional Medical Center, Wilmington, North Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
- Italy (3):
  - Ospedale Civile di Baggiovara, Baggiovara
  - Vincenzo Monaldi Hospital, Napoli
  - Sapienza Università di Roma, Roma
- Spain (2):
  - University Hospital Virgen Macarena - Department of General And Digestive Surgery, Seville
  - Hospital Quirón Salud-Sagrado Corazón, Seville
- United Kingdom (2):
  - University Hospitals Birmingham NHS Foundation Trust - Queen Elizabeth Hospital Birmingham, Birmingham
  - Walsall Manor Hospital, Walsall

IPD SHARING:
Plan to Share IPD: No